CLINICAL TRIAL: NCT02885454
Title: A Phase 1, Open-label Study in Healthy Female Subjects to Investigate the Effects of Odalasvir and AL-335 at Steady-state, Given as Single Agents and in Combination With Simeprevir, on the Single-dose Pharmacokinetics of Ethinylestradiol and Drospirenone
Brief Title: To Evaluate the Effects of Odalasvir and AL-335 With Simeprevir on the Single-Dose Pharmacokinetics of Ethinylestradiol and Drospirenone in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108177; 64294178HPC1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination; adafosbuvir; odalasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OC + AL-335 + ODV + 3-DAA combination (Experimental): Participants will receive single dose of 3 milligram (mg) drospirenone/0.02 mg ethinylestradiol [OC] on Day 1, AL-335 800 mg once daily on Days 5 and 6, a single dose of AL-335 800 mg + a single dose of OC on Day 7, ODV 25 mg once daily on Days 12 to 24, followed by a single dose of ODV 25 mg and a single dose of OC on Day 25, followed by ODV 25 mg + AL-335 800 mg + simeprevir (SMV) 75 mg [3-DAA combination] once daily on Days 26 to 31, followed by a single dose of 3-DAA combination and a single dose of OC on Day 32.
  Interventions: Drug: Drospirenone/ethinylestradiol; Drug: AL-335; Drug: Odalasvir (ODV); Drug: Simeprevir (SMV)

INTERVENTIONS:
Drug: Drospirenone/ethinylestradiol — Each tablet contains 3 mg drospirenone and 0.02 mg ethinylestradiol to be taken orally on Days 1, 6, 25, and 32.
  Other Names: Yaz®
Drug: AL-335 — AL-335 (800 mg) tablet once daily on Days 5-7 and then on Days 26-32 (as a component of 3-DAA combination) to be taken orally.
Drug: Odalasvir (ODV) — ODV 25 mg tablet once daily on Days 12-25 and then on Days 26-32 (as a component of 3-DAA combination) to be taken orally.
Drug: Simeprevir (SMV) — SMV 75 mg capsule as a component of 3-DAA combination to be taken orally on Days 26-32.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state concentrations of odalasvir (ODV), AL-335 and the combination of the 3-direct-acting anti-viral agents (3-DAA) ODV, AL-335, and simeprevir (SMV) on the single-dose pharmacokinetic (PK) of drospirenone and ethinylestradiol in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a female of childbearing potential with a normal menstrual cycle
* Participant must have a body mass index (BMI; weight in kg divided by the square of height in meters) between 18.0 and 30.0 kilogram per square meter (kg/m^2), extremes included, and a body weight not less than 50.0 kilogram (kg)
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Participant must have a negative serum (beta human chorionic gonadotropin [beta- hCG]) pregnancy test at screening
* Participant must have a negative highly sensitive urine pregnancy test at Day -1

Exclusion Criteria:

* Participant is peri- or postmenopausal, or participant with bilateral oophorectomia
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening
* Participant has previously been dosed with simeprevir (SMV), odalasvir (ODV), or AL-335 in more than 3 single dose studies, or a multiple-dose study with SMV, ODV, or AL-335
* Participant with currently active gynecological disorders including, but not limited to, vaginal bleeding without an obvious reason and hyperprolactinemia with or without galactorrhea
* Participant with a past history of: heart arrhythmias (example, extrasystolic rhythms or tachycardia at rest). Isolated extrasystolic beats are not exclusionary; risk factors associated with Torsade de Pointes such as hypokalemia; family history of short/long QT syndrome; sudden unexplained death (including sudden infant death syndrome [SIDS]) in a first-degree relative (that is, sibling, offspring, or biological parent)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Drospirenone | Day 1, 7, 25 and 32: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours postdose
  Cmax is the maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Drospirenone | Day 1, 7, 25 and 32: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Drospirenone | Day 1, 7, 25 and 32: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Maximum Observed Plasma Concentration (Cmax) of Ethinylestradiol | Day 1, 7, 25 and 32: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours postdose
  Cmax is the maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of Ethinylestradiol | Day 1, 7, 25 and 32: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Ethinylestradiol | Day 1, 7, 25 and 32: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 48 and 72 hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Approximately 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States